CLINICAL TRIAL: NCT06291883
Title: Evaluation of KGR Prescriptions in Suppressing COVID-19 Infection.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sheng-Teng Huang (Other)
Responsible Party: Sponsor-Investigator, Sheng-Teng Huang, Attending physician, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CHUH112-REC2-008
Record Dates: First submitted 2024-03-01; First posted 2024-03-04 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Coronavirus Disease 2019; Severe Acute Respiratory Syndrome Coronavirus 2 Infection
Keywords: coronavirus disease 2019; severe acute respiratory syndrome coronavirus 2; Kang Guan Recipe; variants of concern; angiotensin-converting enzyme 2
MeSH Terms: conditions — COVID-19 | interventions — Coal Tar

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treat (Experimental): four packets of concentrated powder per day.
  Interventions: Combination Product: Kang Guan Recipe (Treat)
- Control (Placebo Comparator): four packets of concentrated powder per day.
  Interventions: Combination Product: Kang Guan Recipe (Placebo)

INTERVENTIONS:
Combination Product: Kang Guan Recipe (Treat) — Accurately weigh the Chinese medicinal herbs in the formula by weight, conduct the origin identification of the medicinal materials, and follow the scientific traditional Chinese medicine preparation process. After extraction, concentration, and granulation, package them in aluminum foil, with each package containing 6 grams of concentrated powder.
  Arms: Treat
Combination Product: Kang Guan Recipe (Placebo) — Use 3% Kang Guan Recipe concentrated powder, mix evenly with starch, and package in aluminum foil, with each package containing 6 grams of concentrated powder.
  Arms: Control

SUMMARY:
These studies offer valuable insights into the potential development of KGR as a novel herbal-based preventive and therapeutic strategy against COVID-19.

DETAILED DESCRIPTION:
The ongoing coronavirus disease 2019 (COVID-19) pandemic continues to present challenges despite widespread vaccination efforts, with breakthrough infections remaining a concern. This has led to increased interest in exploring alternative preventive measures, including dietary and natural product-based interventions. Previous studies have demonstrated the potential of herbal medicines in inhibiting viral infections and as therapies for COVID-19. Additionally, research has identified various herbal medicines with inhibitory properties against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, highlighting their potential in combating the virus. Here Researchers found that novel herbal medicine formula Kang Guan Recipe (KGR) is a potent inhibitor against SARS-CoV-2 viral infection. Researchers demonstrated that KGR showed inhibitory activity against variants of concern (VOCs) of SARS-CoV-2 infection. Moreover, they also found that KGR can block the interaction of viral Spike and human angiotensin-converting enzyme 2 (ACE2). Furthermore, Researchers assessed the inhibitory effect of KGR on SARS-CoV-2 viral entry in vivo and observed that serum samples from healthy human subjects exhibited suppressive activity against various SARS-CoV-2 variants after consuming KGR. These studies offer valuable insights into the potential development of KGR as a novel herbal-based preventive and therapeutic strategy against COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged 20-60 with a body weight of over 50 kilograms.
* Individuals who have never been diagnosed with COVID-19 or have recovered from COVID-19 for more than three months.
* No consumption of any traditional Chinese medicine or food containing Chinese medicine within the preceding 36 hours before the experiment.
* Vaccinated individuals who received their vaccine more than three months ago.
* Willingness to undergo venous blood tests (approximately 10 cc of blood to be drawn three times).

Exclusion Criteria:

* History of major internal medical conditions, including diabetes, hypertension, chronic obstructive pulmonary disease (COPD), asthma, abnormal liver function (AST levels exceeding 5 times the normal value), renal dysfunction (eGFR <60), cancer, etc.
* Brain disorders such as trauma, stroke, tumors, epilepsy, or dementia.
* Mental health disorders such as depression, anorexia nervosa, or schizophrenia.
* Pregnant or lactating women. If there is suspicion of pregnancy, a commercial urine pregnancy test will be conducted.
* Smokers, alcoholics, or betel nut addicts.
* Inability to comply with the trial procedures.
* Inability to sign the informed consent form.
* Within three months of a confirmed COVID-19 diagnosis.
* Within three months of receiving a vaccine shot.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Serum Infection rate of pseudocells | Before taking, 2 hours after taking, and 2 hours after taking 24 hours later.
  Collected Blood, centrifuge to obtain serum samples. Each serum sample were diluted and premixed with wild-type or different variants of SARS-CoV-2 spike Vpps for one hours before incubation with 293T-ACE2 cells. After 24 hours of infection, the infection efficiency rate was measured according to luciferase activities.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Teng Huang, MD PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan